CLINICAL TRIAL: NCT04629781
Title: Open-label Dose Escalation Phase 1b Trial of a New Micellar Docetaxel Compound in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Open-label Dose Escalation Phase 1b Trial of a New Micellar Docetaxel Compound in Patients With mCRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: SAKK decided to premature terminate this trial as additional follow-up visits do not further contribute to the efficacy data. This decision does not adversely impact the patients.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 67/20
Record Dates: First submitted 2020-10-22; First posted 2020-11-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer; micellar docetaxel compound; anti-cancer agent; Docecal; Docetaxel

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, single-stage phase 1b trial in patients with mCRPC. A 3+3 design is used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel micellar (Experimental): Trial Treatment with Docetaxel micellar
  Interventions: Drug: Docetaxel micellar

INTERVENTIONS:
Drug: Docetaxel micellar — There will be three dose levels, 1-3, with each level consisting initially of a cohort containing 3 patients. One additional dose level, dose level -1, shall be allowed in the event that dose level 1 is considered too toxic

SUMMARY:
Treatment with polysorbate 80-solved Docetaxel (Taxotere®) is hampered by the requirement to co-administer steroids. Chronic (intermittent) steroids are negatively impacting bone health and have well known immunosuppressive effects. Despite steroid premedication, polysorbate 80-solved Docetaxel (Taxotere®) results in occasional infusion reactions due to the solvent polysorbate 80. Docetaxel micellar is a promising alternative to polysorbate 80-solved Docetaxel (Taxotere) as it avoids the mandatory need for steroid administration pre and post infusion, and thus avoids immunosuppressive and bone-damaging effects.

There is an unmet medical need to develop steroid-free taxane regimens for patients with advanced cancer to avoid the need for steroid administration pre and post infusion (as outlined above). The unique Docetaxel micellar formulation suggests an improved safety profile compared to polysorbate 80-solved Docetaxel (Taxotere®).

DETAILED DESCRIPTION:
Docetaxel, a semi-synthetic analogue of paclitaxel, is one of the most widely used human anti-cancer agents. Docetaxel and paclitaxel belong to a group of cytotoxic agents called taxanes. Docetaxel has been marketed worldwide by Sanofi-Aventis under the trade name Taxotere® and its use is approved for different types of solid tumors. The efficacy of docetaxel has been proven in two different phase 3 trials in metastatic castration resistant prostate cancer (mCRPC) and is a standard of care option for patients with prostate cancer. In Taxotere®, polysorbate 80 is used as surfactant. Fluid retention and hypersensitivity reactions are reported, and the patients are pre-treated with corticosteroids, e.g. dexamethasone, to avoid or at least reduce the frequency and the severity of both hypersensitivity reactions and fluid retention.

Oasmia Pharmaceutical AB (Uppsala, Sweden) has developed a novel formulation of docetaxel (Docetaxel micellar) with N-(all-trans-retinoyl)-L-cysteic acid methyl ester sodium salt (XMeNa) as excipient, thus reducing adverse reactions caused by polysorbate 80. XMeNa forms micelles into which docetaxel can be incorporated thus increasing its aqueous solubility and keeping it dissolved.

Rational Treatment with polysorbate 80-solved Docetaxel (Taxotere) is hampered by the requirement to co-administer steroid pre and post Taxotere infusion. Chronic (intermittent) steroids are hurting bone health and have well known immunosuppressive effects. Despite steroid premedication, polysorbate 80-solved Docetaxel (Taxotere) results in occasional infusion reactions due to the solvent polysorbate 80. The new micellar formulation of docetaxel is a promising alternative to polysorbate 80-solved Docetaxel (Taxotere) as it avoids the mandatory need for steroid administration pre and post infusion, and thus avoids immunosuppressive and bone-damaging effects.

Safety and pharmacokinetics (PK) of Docetaxel micellar have been assessed in 2 clinical studies, but only in breast cancer patients. This is the first clinical trial to assess the safety and tolerability of 3-weekly intravenous Docetaxel micellar infusions in patients with mCRPC.

The primary objective of this study is to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) for Docetaxel micellar in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH GCP E6(R2) regulations before registration and prior to any trial specific procedures.
* Histologically confirmed adenocarcinoma of the prostate
* Metastatic castration resistant, progressive disease as defined as per PCWG3 criteria
* Ongoing concurrent use of GnRH agonist or antagonist is required if the patient has not been surgically castrated
* Measurable or evaluable disease per Recist 1.1 and as per PCWG3
* Patients with treated and stable CNS metastases are eligible, provided they meet the following criteria:

  * No ongoing requirement for corticosteroids as therapy for symptomatic CNS disease; anticonvulsants at a stable dose allowed
  * No stereotactic radiation or whole-brain radiation within 7 days prior to registration,
  * No evidence of progression for at least 4 weeks after completion of CNS-directed therapy as verified by clinical examination and brain imaging (MRI or CT) during the screening period
* Patients with a previously treated malignancy are eligible, when the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low.
* Age ≥ 18 years
* ECOG performance status 0-1
* Adequate bone marrow function: (patient must not have received any growth factor or blood transfusion within 7 days prior to registration): neutrophil count ≥ 1.5 x 109/L , platelet count ≥ 100 x 109/L, hemoglobin ≥ 80 g/L
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease 3.0 x ULN), AST and ALT ≤ 2.5 x ULN
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 (according to CKD-EPI formula)
* Willingness to have a central venous line inserted (PICC or Porth-a-Cath) if not already present.
* Men agree not to donate sperm or to father a child during trial treatment and until 6 months after the last dose of investigational drug. Sexually active patients must agree to have an effective contraception during study treatment and for 6 months after the last dose.

Exclusion Criteria:

* Clinical or radiological evidence of spinal cord compression
* Known predominant small cell or neuroendocrine component on histological diagnosis
* Prior chemotherapy including docetaxel for the treatment of prostate cancer (previous administration of chemotherapy concomitant with ADT is not allowed )
* Prior use of taxane-based chemotherapy for any other previous cancer
* Prior systemic treatment, immunotherapy, hormonal therapy (with the exception of GnRH agonists or antagonists) or investigational agents within 21 days before registration, with the exception of palliative radiotherapy (within 2 weeks)
* Concomitant or within 28 days of registration treatment with any other experimental drug (enrollment in another clinical trial except participation in SAKK 96/12 and/or 63/12]
* Concomitant use of other anti-cancer drugs (other than GnRH agonists or antagonists). Bone-modifying agents (such as bisphosphonates or denosumab) are allowed before study entry and during treatment.
* Patients who have not recovered to CTCAE grade ≤1 from clinically relevant adverse events of prior therapies, except for residual toxicities, such as alopecia, which do not pose an ongoing medical risk.
* Peripheral neuropathy > CTCAE grade 1
* Localized or general edema > CTCAE grade 1
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV; unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), known significant QT-prolongation, uncontrolled hypertension.
* Major surgery within 4 weeks prior to registration
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
* Concomitant or prior use of immunosuppressive medication within 28 days before registration, with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids which must not exceed 10 mg/day of prednisone or a dose equivalent corticosteroid)
* Concomitant treatment with strong CYP3A inducers or inhibitors
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | at the end of Cycle 1 (each cycle is 21 days)
  DLT is defined as the occurrence of any of a set of specified hematological, hepatic, gastro-intestinal, nervous systems disorders, fluid retention or other adverse events (AEs) which:
  * occur during cycle 1 of the trial treatment defined as the DLT monitoring period
  * is considered by the Investigator or the Sponsor to be at least possibly related to the IMP.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | from date of treatment start to date of radiographic progression, or death due to any cause, whichever occurs first, assessed up to 36 months
  rPFS is defined as the time from treatment start to radiographic progression, or death due to any cause, whichever occurs first. The assessment of radiographic disease progression is based on local evaluations.
Time to PSA progression | from date of treatment start to date of PSA progression, or start of a subsequent anticancer treatment, whichever occurs first, assessed up to 36 months
  Time to PSA progression is defined as the time from treatment start to the time point of PSA progression. The PSA progression date is defined as the date of
  * ≥ 25% increase AND ≥ 2 ng/mL increase above the nadir, confirmed by a second value ≥ 3 weeks later, if there is PSA decline from baseline (last PSA measurement before treatment start), or
  * ≥ 25% increase AND ≥ 2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline Time to PSA progression is defined as the time from treatment start to the time point of PSA progression. The PSA progression date is defined as the date of
  * ≥ 25% increase AND ≥ 2 ng/mL increase above the nadir, confirmed by a second value ≥ 3 weeks later, if there is PSA decline from baseline (last PSA measurement before treatment start), or
  * ≥ 25% increase AND ≥ 2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline
PSA response | from date of treatment start to date of end of treatment, assessed up to 30 weeks
  PSA response is defined as a PSA decline of ≥ 50% from baseline measured twice at least 3 weeks apart during treatment.
Partial (PR) or complete (CR) radiological soft tissue response according to RECIST 1.1 | from date of treatment start to date of end of treatment, assessed up to 30 weeks
  Partial (PR) or complete (CR) radiological soft tissue response achieved according to RECIST 1.1 criteria. Patients without any response assessment during trial treatment will be considered as having a non-evaluable response (NE) and thus will be regarded as failure for this endpoint.
Duration of response (DoR) according to RECIST 1.1 | from date of response to date of disease progression according to RECIST 1.1 or death, whichever occurs first, assessed up to 36 months
  DoR is defined as the time from the earliest date of the first documented evidence of complete response (CR) or partial response (PR) until earliest date of disease progression according to RECIST 1.1 or death due to any cause, whichever occurs first.
  Patients not experiencing an event at the time of the analysis, as well as patients starting a subsequent anticancer treatment in the absence of an event, will be censored at the date of their last available tumor assessment before starting a subsequent anticancer treatment, if any.
Adverse Events | From registration until 28 days after last dose of trial treatment
  AEs will be assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Colombo, MD, Study Chair — IOSI, Ospedale San Giovanni, Bellinzona
Locations (3):
- Switzerland (3):
  - IOSI - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital St. Gallen, Sankt Gallen